CLINICAL TRIAL: NCT04297943
Title: The Effectiveness of 3D Printed, Low Temperature Thermoplastic, and Prefabricated Orthoses in the Management of Thumb Carpo-metacarpal Osteoarthritis: A Randomized, Controlled Trial.
Brief Title: Orthotic Management of CMC Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Collaborators: St. Joseph's Healthcare Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115441
Record Dates: First submitted 2020-02-24; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Arthritis Wrist
Keywords: arthritis; orthotics
MeSH Terms: conditions — Arthritis | interventions — Four-Dimensional Computed Tomography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Orthosis (Active Comparator): See summary
  Interventions: Device: Orthosis fabrication; Device: Thermal Sensor Monitoring of Orthosis Use; Diagnostic Test: 4D CT Scan
- Custom Thermoplastic Orthosis (Active Comparator): See summary
  Interventions: Device: Orthosis fabrication; Device: Thermal Sensor Monitoring of Orthosis Use; Diagnostic Test: 4D CT Scan

INTERVENTIONS:
Device: Orthosis fabrication — see summary
Device: Thermal Sensor Monitoring of Orthosis Use — see summary
Diagnostic Test: 4D CT Scan — see summary

SUMMARY:
This study will investigate the effectiveness of 3D printed splints for the treatment of thumb osteoarthritis (CMC OA). Currently, these splints are made by Occupational Therapists and Physical Therapists out of low temperature plastic, and formed on the patient's hand. 3D printed splints involve taking a photographic scan of the hand and creating a digital file of the splint. This is then printed and fit on the patient. This study will compare the effectiveness of these methods of splint fabrication. Our outcomes will include measurements of pain relief, adherence, patient satisfaction, muscle contraction and CT imaging during pinch tasks to measure the ability of these splint types to support the CMC joint.

DETAILED DESCRIPTION:
This study will be prospective, randomized, controlled trial. Patients will be identified for potential inclusion by the surgeons at HULC. The standard of clinical care is for diagnosis of CMC is to perform X-rays of the hand and this is done routinely. Based on these images and clinical evaluation, surgeons will establish a diagnosis of CMC, and provide a grading of severity based on the Eaton/Littler Classification on a referral pad. Eligible participants will then be asked to attend the Clinical Research Laboratory within HULC, where one of the co-investigators listed will present the letter of information and obtain informed consent. Patients who agree to participate will be asked to complete 3 functional outcomes questionnaires (i.e. DASH, PRWHE, and VAS pain scale). Bilateral wrist and thumb range of motion, lateral and tripod pinch strength, and grip strength will also be assessed.

Following the initial assessment, patients will be randomized into one of two groups. Patients will be stratified based on their initial referral by the hand surgeon according to CMC OA severity results to ensure that equal numbers of participants fall into each treatment arm based on the Eaton Classification of their CMC OA. After randomization, patients will attend splinting visit #1 (based on scheduling availability) either the Hand Therapy Department at St. Joseph's Health Care London or Hand Therapy Canada, a private clinic in London. Regardless of group allocation or location of therapy visit, patients will not be charged for their therapy visits or for their splint.

Splinting Visit #1

Group one will be fit with a low temperature custom thermoplastic brace at one of the aforementioned clinic locations and then booked for a follow up appointment in the clinical research laboratory at SJHC two weeks later.

Group two will have their hand placed in a scanner that takes multiple photographs of the hand and reconstructs these photos into a single 3 dimensional computer image. From there, one of the co-investigators (MS) will "draw" the splint, and send to a 3D printer. Patients will come back to a clinic location for fitting, and will then follow up 2 weeks after splint fitting at the clinical research laboratory 2 weeks later.

Regardless of group allocation, each splint will have a temperature sensor placed into the splint. This sensor is similar to a watch battery and collects and records several thousand temperature readings on pre-set intervals. Participants will be told that the the sensor records data on position of the hand in space, but in fact, recording the temperature will provide information about adherence with the splinting program.

CT Scan

Patients undergo a 4D CT scan of bilateral thumb CMC joints. This will include scans at rest, while performing lateral pinch of 2kg, 5kg, and maximum pinch (if greater than 5kg). They will then apply their splint, and these images will be repeated while wearing the splint.

Follow Up Visits

Participants will be asked to wear their splint during most functional activities for 8 weeks, with the goal of wearing their splint for at least half of their waking hours. They will be asked to keep a daily logbook of the amount of time spent in the splint and will keep these records until the 2-month visit. All participants will return to therapy once every 2 weeks. The purpose of these follow up visits will be to download the data from the temperature sensors and to ensure there is no skin irritation or evidence of any skin breakdown from splint use.

2-month visit

At 2 months, participants will be asked to repeat the three functional outcomes questionnaires and will have their ROM and strength re-tested as in visit #1. They will also have a surface EMG recording of their muscle contractions while in the splint. At this point, the sensors will be removed from the splints for final analysis. Patients will also turn in their logbooks of splint usage, and complete a splinting satisfaction questionnaire. They will then attend a second visit to the CT scanner for a repeat imaging session exactly as listed above.

Final Visit

Participants will be call back to the clinic for a final evaluation at 12 months. At this point, all measures will be repeated with the exception of the CT scans.

ELIGIBILITY:
Inclusion Criteria:

All patients with a diagnosis of CMC OA

Exclusion Criteria:

Language barriers Cognitive barriers Previous thumb metacarpal fracture Advanced scapho-trapezial OA

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Disabilities of the Arm Shoulder and Hand Questionnaire. | Initial Visit, at 2 month visit, and at 1 year
  Patient reported outcome measure
Change in Pain | Initial Visit, at 2 month visit, and at 1 year
  VAS scale for pain
4D CT Scan Changes | At enrolment and again 2 months later
  Effectiveness of Orthosis to stabilize CMC while pinching

SECONDARY OUTCOMES:
Adherence | Measured at 2 month visit, with data downloaded biweekly
  Measured via log book and temperature sensors
Orthosis Satisfaction Survey | At 2 month visit and at 1 year
  Assessment of participants satisfaction with orthosis
Change in Pinch strength | Measured in CT scans at enrolment and at 2 month visit
  Pinch gauge measurements

IPD SHARING:
Plan to Share IPD: No